CLINICAL TRIAL: NCT00071448
Title: Basal/Bolus Therapy With Insulin Aspart (NovoLog®) Versus Regular Human Insulin (Novolin® R) or Insulin Lispro (Humalog®) in Combination With NPH: An Open-Label, Randomized, Parallel Group, Multicenter Study in Children and Adolescents With Type 1 Diabetes
Brief Title: Insulin Aspart vs. Insulin Lispro vs. Regular Insulin in Paediatric Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANA-2126
Record Dates: First submitted 2003-10-23; First posted 2003-10-24 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin; Insulin Lispro; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin human
Drug: insulin lispro
Drug: insulin aspart

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to to determine whether insulin aspart can be used effectively and safely in paediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with Type 1 diabetes for at least one year
* HbA1c less than 12%
* Willing to administer at least 3 injections per day
* Willing to perform self monitored blood glucose (SMBG) at least 4 times per day, includes subject and/or parent/guardian, as necessary

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 378 (Actual)
Dates: Start 2002-06; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin A1c)

SECONDARY OUTCOMES:
FPG (fasting plasma glucose)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (67):
- United States (67):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Mobile, Alabama
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Loma Linda, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Englewood, Colorado
  - Novo Nordisk Investigational Site, Hartford, Connecticut
  - Novo Nordisk Investigational Site, New Haven, Connecticut
  - Novo Nordisk Investigational Site, Gainesville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Pensacola, Florida
  - Novo Nordisk Investigational Site, Tallahassee, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Baton Rouge, Louisiana
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Worcester, Massachusetts
  - Novo Nordisk Investigational Site, Ann Arbor, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Rochester, Minnesota
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Hackensack, New Jersey
  - Novo Nordisk Investigational Site, Morristown, New Jersey
  - Novo Nordisk Investigational Site, Paterson, New Jersey
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, Mineola, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Akron, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Danville, Pennsylvania
  - Novo Nordisk Investigational Site, Erie, Pennsylvania
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Columbia, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Lackland City, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Temple, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Morgantown, West Virginia
  - Novo Nordisk Investigational Site, Madison, Wisconsin

REFERENCES:
- [Result] Arslanian S, Foster C, Wright N, Stender S, Hu P, Hale P, Hale D. Comparison of Insulin Aspart, Regular Insulin, and Insulin Lispro in Basal Bolus Therapy with NPH To Treat Pediatric Patients with Type 1 Diabetes Mellitus. Diabetes 2005; 54 ((suppl 1)): A517 [Abstract 2150-PO]
- [Result] Arslanian S, Foster C, Wright NM, Stender S, Hale P, Hale D. Insulin apart compared to regular insulin and insulin lispro in basal bolus therapy with NPH to treat pediatric patients with type 1 diabetes mellitus. EASD 2005 2005; 48(Suppl. 1): A327
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com